CLINICAL TRIAL: NCT02475577
Title: A Prospective Randomized Controlled Trial to Determine Return on Investment in a Tablet/Smartphone-based Heart Failure Remote Monitoring Program
Brief Title: Determine Return on Investment in Heart Failure Remote Monitoring Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NCH Healthcare System, Inc. dba Naples Comprehensive Health and dba NCH (Other)
Collaborators: Welch Allyn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-001
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
Keywords: telemedicine; heart failure; home blood pressure monitoring
MeSH Terms: conditions — Heart Failure | interventions — Blood Pressure Monitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Control: Peripherals with HealthInterlink technology will record and transmit data, without intervention. Subject is able to view graphed data, bring the HealthInterlink tablet/smartphone to the physician's office and share data with family/other caregiver.
  Interventions: Device: Peripherals with HealthInterlink technology
- Intervention 1 (Experimental): Intervention 1: Peripherals with HealthInterlink technology will record and transmit data and send out-of-range data (Red) alerts to subject via HealthInterlink tablet/smartphone and also text/email to family/other caregiver, and nonconformity (Blue) alerts to subject's personal text/email and also text/email to family/other caregiver.
  Interventions: Device: Peripherals with HealthInterlink technology
- Intervention 2 (Experimental): Intervention 2: Peripherals with HealthInterlink technology will record and transmit data and send out-of-range data (Red) alerts to subject via HealthInterlink tablet/smartphone and also text/email to family/other caregiver, and nonconformity (Blue) alerts to subject's personal text/email and also text/email to family/other caregiver, and a call will be placed by the nurse research assistant to study subject (on Blue alerts) or study subject's healthcare professional (on Red alerts). The physicians will have access to the subject's data on a web-based program.
  Interventions: Device: Peripherals with HealthInterlink technology

INTERVENTIONS:
Device: Peripherals with HealthInterlink technology — home remote monitoring
  Other Names: Welch Allyn; Blood Pressure monitor; Weight Scale; Pulse Oximeter; tablet/smartphone-based technology

SUMMARY:
The study will test a hypothesis that the remote monitoring with text and email alerts sent to study subject and optional family/other caregiver (Intervention 1) will have a higher return on investment compared to remote monitoring with nurse researcher follow-up telephone communication to study subject (on Blue alerts) or study subject's healthcare professional (on Red alerts) (Intervention 2) and self-monitoring without intervention (Control).

DETAILED DESCRIPTION:
The objective of this remote monitoring study is to evaluate return on investment and end-user clinical outcomes associated with the use of self-monitoring peripherals and tablet/smartphone-based Welch Allyn HealthInterlink technology without intervention (Control), HealthInterlink remote monitoring with text and email alerts sent to study subject and optional family/other caregiver (Intervention 1), and HealthInterlink remote monitoring with nurse research assistant follow-up telephone communication to study subject (on Blue alerts) or study subject's healthcare professional (on Red alerts) (Intervention 2 added to Intervention 1).

ELIGIBILITY:
Inclusion Criteria:

* Absence of significant vision, hearing, or other communication deficits
* English speaking;
* Capable and willing to give informed consent;
* Participated in the in-patient heart failure class within the last three months. Acceptable candidate for elective, non-emergent, remote monitoring as determined by ordering physician;
* Living in a private home;
* Hospital admission for Heart Failure or decompensation in the previous 12 months
* New York Heart Association (NYHA) classes II-IV, as assigned by the nurse researcher, trained by a cardiologist
* Cardiac aetiology: ischaemic, idiopathic, hypertensive, or valvular
* Left ventricular ejection fraction <40% s an index of systolic dysfunction, combined or not with a left ventricular filling pattern supporting the presence of diastolic dysfunction, according to the American College of Cardiology/American Heart Association Guidelines for chronic heart failure.

or

* NYHA class II-III who had an ejection fraction >40% and evidence of diastolic left ventricular dysfunction.
* Optional subject with a diagnosis of diabetes (indicated by HbA1c >7).

Exclusion Criteria:

* Currently involved in other investigational clinical trials (unless permission is granted by other study PI);
* Females who are pregnant, planning to become pregnant within 3 months, or lactating;
* Requirement for emergent placement other than private home (subject's condition would be compromised if there is a delay in placement).
* Myocardial infarction, revascularization or Implantable Cardioverter Defibrillator (ICD) implantation in the previous 6 months angina or objective myocardial ischaemia requiring future revascularization implanted ventricular or atrial pacemaker (except dual chamber ICD pacemakers with good sinus activity);
* End-stage heart failure requiring regular inotropic drug infusions;
* Chronic renal failure requiring dialysis treatment and
* Unstable angina.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with unplanned re- hospitalization (heart failure-related and other hospitalization) | 31 days
  31 days post discharge with a heart failure-related hospital re-hospitalization.

SECONDARY OUTCOMES:
Communication with healthcare provider or emergency department | 31 days
  Communication that resulted in unplanned healthcare provider office visits or visit to emergency department
Number of non-conformity issues | 31 days
  Number of non-conformity telephone reminder texts, emails, and/or calls.
Health-related quality of life Questionnaire | 31 days
  Health-related quality of life
Subject satisfaction Questionnaire | 31 days
  Subject satisfaction for peripherals and HealthInterlink tablet/ smartphone judged to be reliable and robust, ease of use, time to complete testing and questionnaire, benefit that promoted better health
Physician satisfaction Questionnaire | 31 days
  Physician satisfaction for peripherals and HealthInterlink tablet/ smartphone judged to be reliable and robust, ease of use of software, benefit that promoted better communication with subject.
Cost of system and intervention per subjects | 31 days
  Economic viability of remote monitoring program based on daily cost of system and intervention per subjects in comparison with control and treatment groups.

OTHER OUTCOMES:
Number and type of incidents | 31 days
  Number and type of incident based on predefined criteria from the remote monitoring data (clinical signs and symptoms related to worsening of cardiac insufficiency or to its complications).
Subject attrition | 31 days
  Rate of subjects discontinuing the study due to Patient Request, Patient Complaint, Patient Transferred to higher level of care (ACLF, SNF), Patient Hospitalized, Physician Request Monitoring No Longer Needed (Resolution of Disease Process, Change in Treatment), Physician Complaint, Patient Expired, Patient all-cause mortality or Without other identifiable cause.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Morrison, PhD, Principal Investigator — NCH Healthcare System Inc
Locations (1):
- NCH Healthcare System, Naples, Florida, United States

REFERENCES:
- See also: Healthcare system web site — http://nchmd.org